CLINICAL TRIAL: NCT02605993
Title: A Phase 2, Open-label, Multiple Ascending Dose Study to Evaluate the Efficacy, Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of ALXN1210 Administered Intravenously to Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Open-label, Multiple Ascending Dose Study of Ravulizumab (ALXN1210) in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-201; 2015-002674-20 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH
Keywords: complement inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): During the Treatment Period, participants were administered ravulizumab 1400 milligram (mg) on Day 1, ravulizumab 1000 mg on Day 15 and Day 29, and then ravulizumab 1000 mg every 4 weeks for 7 doses.
  In the Extension Period, participants initially continued to receive their dose. During the second year of the study, participants were administered weight-based doses of ravulizumab every 8 weeks for up to 5 years: 3000 mg for participants weighing 40 to less than 60 kilograms (kg), 3300 mg for participants weighing 60 to less than 100 kg, and 3600 mg for participants weighing 100 kg or more.
  Interventions: Biological: Ravulizumab
- Cohort 2 (Experimental): During the Treatment Period, participants were administered ravulizumab 2000 mg on Day 1, ravulizumab 1600 mg on Day 22 and Day 43, and then ravulizumab 1600 mg every 6 weeks for 4 doses.
  In the Extension Period, participants initially continued to receive their dose. During the second year of the study, participants were administered weight-based doses of ravulizumab every 8 weeks for up to 5 years: 3000 mg for participants weighing 40 to less than 60 kg, 3300 mg for participants weighing 60 to less than 100 kg, and 3600 mg for participants weighing 100 kg or more.
  Interventions: Biological: Ravulizumab
- Cohort 3 (Experimental): During the Treatment Period, participants were administered ravulizumab 1600 mg on Day 1 and Day 15, ravulizumab 2400 mg on Day 29, and then ravulizumab 2400 mg every 8 weeks for 3 doses.
  In the Extension Period, participants initially continued to receive their dose. During the second year of the study, participants were administered weight-based doses of ravulizumab every 8 weeks for up to 5 years: 3000 mg for participants weighing 40 to less than 60 kg, 3300 mg for participants weighing 60 to less than 100 kg, and 3600 mg for participants weighing 100 kg or more.
  Interventions: Biological: Ravulizumab
- Cohort 4 (Experimental): During the Treatment Period, participants were administered ravulizumab 3000 mg on Day 1, ravulizumab 5400 mg on Day 29, and then ravulizumab 5400 mg every 12 weeks for 2 doses.
  During the Extension Period, participants were administered ravulizumab 5400 mg every 12 weeks for up to 5 years.
  Interventions: Biological: Ravulizumab

INTERVENTIONS:
Biological: Ravulizumab — All treatments were given as IV infusions.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and efficacy of multiple intravenous (IV) doses of ravulizumab administered to complement inhibitor treatment-naïve participants with PNH.

DETAILED DESCRIPTION:
The study consisted of a screening period of up to 30 days and a Treatment Period of up to 253 days for Cohorts 1-3 and 281 days for Cohort 4. After completion of the Treatment Period, all participants had the opportunity to enter the Extension Period, wherein participants continue to receive ravulizumab for up to 5 years. The first dose in the Extension Period occurred on Day 253 for Cohorts 1-3 and on Day 281 for Cohort 4.

The data presented includes the Primary Completion date of the study for the Treatment Period. The results for the Extension Period will be reported after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. PNH diagnosis confirmed by documented high-sensitivity flow cytometry
3. Documented meningococcal vaccination not more than 3 years prior to dosing
4. Female participants of childbearing potential were to use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.
5. Willing and able to give written informed consent and comply with the study visit schedule

Exclusion Criteria:

1. Treatment with a complement inhibitor at any time
2. Female participants who are planning to become pregnant, or are pregnant, breastfeeding or who had a positive pregnancy test at screening or Day 1
3. Participation in an interventional clinical study within 30 days before initiation of dosing on Day 1, or use of any experimental therapy within 30 days prior to dosing on Day 1, or within 5 half-lives of the investigational product, whichever was greater
4. History of allergy to any drug, allergen, excipients of ravulizumab or known allergy to Chinese hamster ovary cell proteins
5. Inability to comply with study requirements
6. History of any clinically significant cardiac, hepatic, immunologic, pulmonary, or rheumatoid disease that, in the Investigator's judgment, would preclude participation
7. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the participant unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Clinical Trial Site, Toronto, Ontario, Canada
- France (3):
  - Clinical Trial Site, Lyon, Pierre-Bénite
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Paris
- Germany (3):
  - Clinical Trial Site, Ulm, Baden-Wurttemberg
  - Clinical Trial Site, Aachen, North Rhine-Westphalia
  - Clinical Trial Site, Essen, North Rhine-Westphalia
- Clinical Trial Site, Seoul, South Korea
- Spain (4):
  - Clinical Trial Site, Badalona, Barcelona
  - Clinical Trial Site, Majadahonda, Madrid
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
- Clinical Trial Site, Taipei, Taiwan
- United Kingdom (2):
  - Clinical Trial Site, Leeds, West Yorkshire
  - Clinical Trial Site, London

REFERENCES:
- [Derived] Roth A, Rottinghaus ST, Hill A, Bachman ES, Kim JS, Schrezenmeier H, Terriou L, Urbano-Ispizua A, Wells RA, Jang JH, Kulasekararaj AG, Szer J, Aguzzi R, Damokosh AI, Shafner L, Lee JW. Ravulizumab (ALXN1210) in patients with paroxysmal nocturnal hemoglobinuria: results of 2 phase 1b/2 studies. Blood Adv. 2018 Sep 11;2(17):2176-2185. doi: 10.1182/bloodadvances.2018020644. PMID 30171081

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: During the Treatment Period, participants were administered ravulizumab 1400 milligrams (mg) on Day 1, ravulizumab 1000 mg on Day 15 and Day 29, and then ravulizumab 1000 mg every 4 weeks for 7 doses. In the Extension Period, participants initially continued to receive their dose. During the second year of the study, participants were administered weight-based doses of ravulizumab every 8 weeks for up to 5 years: 3000 mg for participants weighing 40 to less than 60 kilograms (kg), 3300 mg for participants weighing 60 to less than 100 kg, and 3600 mg for participants weighing 100 kg or more.
Period: Treatment Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 | 6 | 7 | 7
Received at Least 1 Dose of Study Drug | 6 | 6 | 7 | 7
Completed | 6 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 | 6 | 7 | 7
Received at Least 1 Dose of Study Drug | 6 | 6 | 7 | 7
Completed (Extension Period ongoing) | 6 | 6 | 6 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Participant underwent bone marrow transplantation due to chronic myelomonocytic leukemia | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set: All participants who received at least 1 dose of ravulizumab.
Groups:
- Cohort 1: During the Treatment Period, participants were administered ravulizumab 1400 mg on Day 1, ravulizumab 1000 mg on Day 15 and Day 29, and then ravulizumab 1000 mg every 4 weeks for 7 doses. In the Extension Period, participants initially continued to receive their dose. During the second year of the study, participants were administered weight-based doses of ravulizumab every 8 weeks for up to 5 years: 3000 mg for participants weighing 40 to less than 60 kg, 3300 mg for participants weighing 60 to less than 100 kg, and 3600 mg for participants weighing 100 kg or more.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first infusion of study drug.
  years | 43.1 (14.57) | 48.6 (23.48) | 37.3 (14.03) | 48.5 (13.43) | 44.3 (16.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 6
  Male | 4 | 5 | 6 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 7 | 7 | 22
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 5 | 4 | 3 | 3 | 15
  Asian | 0 | 0 | 4 | 3 | 7
  Not Reported | 1 | 2 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 1 | 1
Lactate Dehydrogenase (LDH) Levels [Mean (Standard Deviation); unit: units/liter (U/L)] | 1026.88 (547.843) | 1223.55 (149.693) | 2127.57 (815.875) | 2142.24 (366.511) | 1668.90 (724.341)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change In LDH Levels From Baseline To Day 253 And Day 281
Description: The percent change in LDH levels was assessed from Baseline to Day 253 for Cohorts 1 to 4 and from Baseline to Day 281 for Cohort 4 only.
Time Frame: Baseline, Day 253 (Cohorts 1 to 4) and Day 281 (Cohort 4)
Population: Full Analysis Set: Participants in the safety set with a Baseline and at least 1 LDH measurement after first dose of ravulizumab. Data summarized only for participants with data at Baseline and the specified time point. Last observation carried forward (LOCF) was used for participants with a missing Day 253 or Day 281 assessment.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Percent Change
  Day 253 | -72.85 (12.082) | -78.12 (6.635) | -84.96 (4.423) | -87.63 (6.923)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 281 |  |  |  | -89.89 (2.885)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; Statistical Analysis presented is of Cohorts 1 to 4 combined at Day 253. A sample size of 20 participants from the combined cohorts was required to provide approximately 95% power to detect a mean paired difference in LDH from Baseline of -40% at Day 253 for Cohorts 1 to 4, with an estimated standard deviation (SD) of 45%. This was based on a 2-sided paired t-test, with 5% type I error rate. To account for a possible 15% dropout rate, up to 26 participants were enrolled; Test type: Other; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — Hypothesis testing was performed at the 0.05 level of significance. P-value tested whether the percent changes differed from 0 for the combined cohorts
Statistical Analysis 2: Comparison: Cohort 4; Statistical Analysis presented is of Cohort 4 at Day 281. A sample size of 20 participants from the combined cohorts was required to provide approximately 95% power to detect a mean paired difference in LDH from Baseline of -40% at Day 281 for Cohort 4 only, with an estimated SD of 45%. This was based on a 2-sided paired t-test, with 5% type I error rate. To account for a possible 15% dropout rate, up to 26 participants were enrolled; Test type: Other; p < 0.0001, MMRM — Hypothesis testing was performed at the 0.05 level of significance. P-value tested whether the percent changes differed from 0

2. Secondary Outcome: Percent Change In Free Hemoglobin Levels From Baseline To Day 253 And Day 281
Description: The percent change in free hemoglobin levels was assessed from Baseline to Day 253 for Cohorts 1 to 4 and from Baseline to Day 281 for Cohort 4 only.
Time Frame: Baseline, Day 253 (Cohorts 1 to 4) and Day 281 (Cohort 4)
Population: Full Analysis Set: Participants in the safety set with a Baseline and at least 1 LDH measurement after first dose of ravulizumab. Data summarized only for participants with data at Baseline and the specified time point. LOCF was used for participants with a missing Day 253 or Day 281 assessment.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Percent Change
  Day 253 | 14.07 (124.755) | -12.32 (57.213) | -22.14 (94.388) | -40.80 (27.474)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 281 |  |  |  | -45.64 (28.938)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; Statistical Analysis presented is of Cohorts 1 to 4 combined at Day 253; Test type: Other; p = 0.0214, MMRM — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 4; Statistical Analysis presented is of Cohort 4 at Day 281; Test type: Other; p = 0.0313, MMRM — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percent Change In Haptoglobin Levels From Baseline To Day 253 And Day 281
Description: The percent change in haptoglobin levels was assessed from Baseline to Day 253 for Cohorts 1 to 4 and from Baseline to Day 281 for Cohort 4 only.
Time Frame: Baseline, Day 253 (Cohorts 1 to 4) and Day 281 (Cohort 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Percent Change
  Day 253 | 21.67 (53.072) | 81.67 (200.042) | 4.29 (11.339) | 34.29 (74.578)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 281 |  |  |  | 27.14 (56.188)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; tatistical Analysis presented is of Cohorts 1 to 4 combined at Day 253; Test type: Other; p = 0.0625, MMRM — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 4; Hypothesis testing was performed at the 0.05 level of significance. P-value tested whether the percent changes differed from 0 for the combined cohorts; Test type: Other — MMRM; p = 0.5000, MMRM — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percent Change In Reticulocyte/Erythrocyte Count From Baseline To Day 253 And Day 281
Description: The percent change in reticulocyte/erythrocyte count levels was assessed from Baseline to Day 253 for Cohorts 1 to 4 and from Baseline to Day 281 for Cohort 4 only.
Time Frame: Baseline, Day 253 (Cohorts 1 to 4) and Day 281 (Cohort 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Percent Change
  Day 253 | -1.27 (43.019) | -5.05 (35.691) | 10.46 (59.510) | 14.66 (81.390)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Day 281 |  |  |  | -4.66 (68.502)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; Statistical Analysis presented is of Cohorts 1 to 4 combined at Day 253; Test type: Other; p = 0.4871, MMRM — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 4; Statistical Analysis presented is of Cohort 4 at Day 281; Test type: Other; p = 0.4688, MMRM — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Percent Change In PNH RBC Types II And III Clone Size From Baseline To Day 253
Description: The percent change in paroxysmal nocturnal hemoglobinuria (PNH) red blood cell (RBC), summed types II and III, clone size levels were assessed from Baseline to Day 253 for Cohorts 1 to 4.
Time Frame: Baseline, Day 253 (Cohorts 1 to 4)
Population: Full Analysis Set: Participants in the safety set with a Baseline and at least 1 LDH measurement after first dose of ravulizumab. Data summarized only for participants with data at Baseline and the specified time point. LOCF was used for participants with a missing Day 253 assessment.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Percent Change | 6.65 (24.101) | 5.47 (21.940) | 54.14 (98.713) | 88.21 (138.290)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; Statistical Analysis presented is of Cohorts 1 to 4 combined at Day 253; Test type: Other; p = 0.0023, MMRM — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Change In D-dimer From Baseline To Day 253 And Day 281
Description: The percent change in D-dimer levels were assessed from Baseline to Day 253 for Cohorts 1 to 4 and from Baseline to Day 281 for Cohort 4 only.
Time Frame: Baseline to Day 253 (Cohorts 1 to 4) and Day 281 (Cohort 4)
Population: Full Analysis Set: Participants in the safety set with a Baseline and at least 1 LDH measurement after first dose of ravulizumab. Data summarized only for participants with data at Baseline and the specified time point. LOCF is used for participants with a missing Day 253 or Day 281 assessment.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 6
Percent Change
  Day 253 | -24.80 (32.436) | -29.47 (26.547) | -10.90 (41.032) | -16.08 (34.783)
  Day 281: number analyzed (Participants) | 0 | 0 | 0 | 6
  Day 281 |  |  |  | -27.05 (27.663)
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 4; Statistical Analysis presented is of Cohorts 1 to 4 combined at Day 253; Test type: Other; p = 0.0029, MMRM — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 4; Statistical Analysis presented is of Cohort 4 at Day 281; Test type: Other; p = 0.1250, MMRM — [p-value comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change In Clinical Manifestations Of PNH From Baseline To Day 253 And Day 281
Description: Clinical manifestations were assessed from Baseline to Day 253 for Cohorts 1 to 3 and from Baseline to Day 281 for Cohort 4 only. Clinical manifestations were defined as fatigue, abdominal pain, dyspnea, dysphagia, chest pain, and erectile dysfunction (male participants only). Improvement was defined as present at Baseline and absent at Day endpoint. Worsening was defined as absent at Baseline and present at Day endpoint. No Change was defined as no change from Baseline and time point of endpoint.
Time Frame: Baseline, Day 253 (Cohorts 1 to 3) and Day 281 (Cohort 4)
Population: Full Analysis Set: Participants in the safety set with a Baseline and at least 1 LDH measurement after first dose of ravulizumab. Data summarized only for participants with data at Baseline and the specified time point. LOCF is used for participants with a missing Day 253 or Day 281 assessment. Erectile dysfunction affects only male participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 6 | 7 | 7
Participants
  Fatigue at Day 253: Improved from Baseline | 4 | 2 | 3 | 3
  Fatigue at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Fatigue at Day 253: No Change | 2 | 4 | 4 | 4
  Fatigue at Day 253: Not Applicable | 0 | 0 | 0 | 0
  Fatigue at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Fatigue at Day 281: Improved from Baseline |  |  |  | 4
  Fatigue at Day 281: Worsened from Baseline |  |  |  | 0
  Fatigue at Day 281: No Change |  |  |  | 3
  Fatigue at Day 281: Not Applicable |  |  |  | 0
  Abdominal Pain at Day 253: Improved from Baseline | 1 | 1 | 1 | 0
  Abdominal Pain at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Abdominal Pain at Day 253: No Change | 5 | 5 | 6 | 7
  Abdominal Pain at Day 253: Not Applicable | 0 | 0 | 0 | 0
  Abdominal Pain at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Abdominal Pain at Day 281: Improved from Baseline |  |  |  | 0
  Abdominal Pain at Day 281: Worsened from Baseline |  |  |  | 0
  Abdominal Pain at Day 281: No Change |  |  |  | 7
  Abdominal Pain at Day 281: Not Applicable |  |  |  | 0
  Dyspnea at Day 253: Improved from Baseline | 1 | 1 | 4 | 2
  Dyspnea at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Dyspnea at Day 253: No Change | 5 | 5 | 3 | 5
  Dyspnea at Day 253: Not Applicable | 0 | 0 | 0 | 0
  Dyspnea at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Dyspnea at Day 281: Improved from Baseline |  |  |  | 2
  Dyspnea at Day 281: Worsened from Baseline |  |  |  | 0
  Dyspnea at Day 281: No Change |  |  |  | 5
  Dyspnea at Day 281: Not Applicable |  |  |  | 0
  Dysphagia at Day 253: Improved from Baseline | 0 | 1 | 1 | 1
  Dysphagia at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Dysphagia at Day 253: No Change | 6 | 5 | 6 | 6
  Dysphagia at Day 253: Not Applicable | 0 | 0 | 0 | 0
  Dysphagia at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Dysphagia at Day 281: Improved from Baseline |  |  |  | 1
  Dysphagia at Day 281: Worsened from Baseline |  |  |  | 0
  Dysphagia at Day 281: No Change |  |  |  | 6
  Dysphagia at Day 281: Not Applicable |  |  |  | 0
  Chest Pain at Day 253: Improved from Baseline | 1 | 0 | 2 | 0
  Chest Pain at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Chest Pain at Day 253: No Change | 5 | 6 | 5 | 7
  Chest Pain at Day 253: Not Applicable | 0 | 0 | 0 | 0
  Chest Pain at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Chest Pain at Day 281: Improved from Baseline |  |  |  | 0
  Chest Pain at Day 281: Worsened from Baseline |  |  |  | 0
  Chest Pain at Day 281: No Change |  |  |  | 7
  Chest Pain at Day 281: Not Applicable |  |  |  | 0
  Erectile Dysfunction at Day 253: Improved from Baseline | 2 | 0 | 1 | 1
  Erectile Dysfunction at Day 253: Worsened from Baseline | 0 | 0 | 0 | 0
  Erectile Dysfunction at Day 253: No Change | 2 | 5 | 5 | 4
  Erectile Dysfunction at Day 253: Not Applicable | 2 | 1 | 1 | 2
  Erectile Dysfunction at Day 281: number analyzed (Participants) | 0 | 0 | 0 | 7
  Erectile Dysfunction at Day 281: Improved from Baseline |  |  |  | 1
  Erectile Dysfunction at Day 281: Worsened from Baseline |  |  |  | 0
  Erectile Dysfunction at Day 281: No Change |  |  |  | 4
  Erectile Dysfunction at Day 281: Not Applicable |  |  |  | 2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously from Screening to Day 253 (for Cohorts 1, 2, and 3) and Day 281 (for Cohort 4) (Treatment Period) and up to Day 2157 (Extension Period).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 4/7 | 1/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Meningococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gonococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=7) | Cohort 4 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Chest pain (General disorders) | 2 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Pain (General disorders) | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 5 | 4
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 2
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 3 | 5 | 4 | 3
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 2 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02605993/Prot_002.pdf
  • Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02605993/SAP_003.pdf